CLINICAL TRIAL: NCT03338075
Title: Fractionated Stereotactic Radiotherapy Combined With Temozolomide for Large Brain Metastases: a Propensity-matched Study
Brief Title: FSRT Combined With TMZ for Large BMs: a PSM Study
Status: Completed | Type: Observational
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jianping Xiao, Dr, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: CH-H&N-004
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Brain Metastases; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Brain Neoplasms | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRT group: patients with brain metastases of more than 6 cc and treated with fractionated stereotactic radiotherapy plus concomitant Temozolomide.
  Interventions: Radiation: fractionated stereotactic radiotherapy
- RT group: patients with brain metastases of more than 6 cc and treated with fractionated stereotactic radiotherapy alone.
  Interventions: Radiation: fractionated stereotactic radiotherapy

INTERVENTIONS:
Radiation: fractionated stereotactic radiotherapy — The regular prescription doses were 52 Gy in 13 fractions or 52.5 Gy in 15 fractions.
  Other Names: drugs

SUMMARY:
A propensity- matched study was conducted to investigate the feasibility and safety of adding temozolomide to hypofractionated stereotactic radiotherapy for large brain metastases.

DETAILED DESCRIPTION:
A previous single arm phase II trial of our institution has shown that HFSRT combined with concurrent TMZ was safe and efficient for patients with BMs of ≥ 6cc in volume. The 1-year local control and overall survival rate was better than the results of a retrospective study using HFSRT alone in treating BMs of ≥ 3cm in diameter. Thus, we hypothesized that adding TMZ to HFSRT should translate to substantive benefits in clinical outcomes compared to HFSRT alone. Propensity score matching method was adopted to decrease potential bias in this retrospective study.

ELIGIBILITY:
Inclusion Criteria:

* (1) primary tumor was pathologically diagnosed and brain metastases were confirmed by gadolinium-enhanced magnetic resonance imaging (MRI) ; (2) age 18 years or older (3) KPS ≥60, or KPS ≥50 but symptomatically caused by BMs; (4) the large lesions haven't treated with surgery or SRT.

Exclusion Criteria:

* (1) KPS <60 but not caused by BMs; (2) the large lesions have been treated with surgery or SRT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with large brain metastases of more than 6 cc.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Local tumor control rate (LTCR) | 3 months after radiation
  the control rate of treated lesions

SECONDARY OUTCOMES:
Intracranial progression- free survival (IPFS) | up to 1 year
  the interval from the beginning of radiation to any intracranial progression
Local recurrence- free survival (LRFS) | up to 1 year
  the time from the beginning of radiation to local faliure.
Overall survival (OS) | up to 3 years
  the time from the beginning of radiation to follow-up or death
Progression- free survival (PFS) | up to 1 year
  the interval from the beginning of HFSRT to any progression of tumor.
Brain metastasis-specific survival (BMSS) | up to 1 year
  the internal from the beginning of radiation to death that caused by brain metastases.

CONTACTS AND LOCATIONS:
Overall Officials: Jianping Xiao, Dr, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: No